CLINICAL TRIAL: NCT03100539
Title: Trial Outcomes for Massage: Caregiver-Assisted vs. Therapist-Treated (TOMCATT)
Brief Title: Trial Outcomes for Massage: Caregiver-Assisted vs. Therapist-Treated
Acronym: TOMCATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 15-333
Record Dates: First submitted 2017-03-06; First posted 2017-04-04 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain; Chronic Pain; Pain; Arthritis; Musculoskeletal Pain; Osteoarthritis
Keywords: Massage; Fascia
MeSH Terms: conditions — Neck Pain; Chronic Pain; Pain; Arthritis; Musculoskeletal Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Therapist treated massage (TT-M) (Experimental): Participants randomized to the therapist-treated massage (TT-M) arm will receive a standardized Swedish massage protocol tailored to chronic neck pain. Massage sessions will involve a maximum of 60 minutes of hands-on, table time and occur twice a week (a frequency which balances practicality and efficacy) for 3 months.
  Interventions: Other: Therapist treated massage
- Wait list control (WL-C) (No Intervention): Participants in the waitlist control will be instructed to continue their medical care as normal and to not begin any massage treatment during the 6 months of the study. At the competition of the final 6 month outcome, participants in the control arm will be eligible to attend a caregiver training session and receive a complementary massage session from a TOMCATT study therapist.
- Care ally assisted massage (CA-M) (Experimental): CA-M consisted of in-person training for veteran/care-ally dyads to learn a standardized 30-minue massage routine, instructional DVD, and printed treatment manual. Participants were to complete three care ally-assisted massage sessions weekly for 12-weeks.
  Interventions: Other: Care ally assisted massage

INTERVENTIONS:
Other: Therapist treated massage — Participants randomized to the therapist-treated massage (TT-M) arm will receive a standardized Swedish massage protocol tailored to chronic neck pain. Massage sessions will involve a maximum of 60 minutes of hands-on, table time and occur twice a week (a frequency which balances practicality and efficacy) for 3 months.
  Other Names: TT-M
  Arms: Therapist treated massage (TT-M)
Other: Care ally assisted massage — CA-M consisted of in-person training for veteran/care-ally dyads to learn a standardized 30-minue massage routine, instructional DVD, and printed treatment manual. Participants were to complete three care ally-assisted massage sessions weekly for 12-weeks.
  Other Names: CA-M
  Arms: Care ally assisted massage (CA-M)

SUMMARY:
Given the modest effectiveness of current treatments and the burden chronic neck pain places on Veterans, the investigators' research proposal is significant in several regards. First, Trial Outcomes for Massage: Caregiver-Assisted vs. Therapist-Treated (TOMCATT) Study directly addresses a high priority area for the VA and is well aligned with the VHA Pain Management Strategy and VHA Pain Management Directive 2009-053. Second, because previous massage studies have included relatively small sample sizes, this trial will provide information vital to fill an evidence vacuum regarding effectiveness of a massage treatments for chronic neck pain. Third, TOMCATT will extend the current understanding of non-pharmacological treatments. Fourth, if the study hypotheses are corroborated massage may emerge as an effective, safe, affordable, sustainable, and accessible treatment for Veterans.

DETAILED DESCRIPTION:
Background: Neck pain is the fourth leading cause of disability in the US, after back pain, depression, and joint pain, and accounts for more than 10 million medical visits per year. Conventional treatments (medications, physical therapy) are widely used for chronic neck pain, yet have modest effectiveness and may carry risks, such as the toxicities associated with non-steroidal anti-inflammatory drugs (NSAIDs) and opioids. As a result many patients live with chronic, often debilitating, pain. Patients unable to find relief frequently turn to complementary health approaches. Complementary therapies are exceptionally popular among Veterans; 82% reported use of at least one complementary therapy and nearly all (99%) were willing to try massage for pain relief. Neck pain is the second most common reason for using a complementary therapy, with massage used for neck pain more commonly than all other complementary therapies except chiropractic care. Of all complementary approaches, massage was the most preferred by Veterans. In a national survey, almost two-thirds (61%) of individuals with neck pain who used both complementary and conventional treatments perceived complementary to be more helpful, whereas only 6% perceived conventional treatments to be better.

Objectives: The Trial Outcomes for Massage: Caregiver-Assisted vs. Therapist-Treated (TOMCATT) Study is a 2-arm, parallel group, randomized clinical trial that will last 6 months. The TOMCATT Study will target 264 Veterans with chronic neck pain and will compare therapist-treated massage to a waitlist control arm on primary, secondary, and exploratory outcomes. There was previously an additional group staff randomized 102 Veterans and their Care Allies to, but are no longer randomizing into this group.

Methods: This study sample will include 264 Veterans with chronic neck pain. Patients from the 5 primary care clinics at the Roudebush VA Medical Center (RVAMC) and 3 community based outpatient clinics (Terre Haute, Martinsville, and Bloomington) will be recruited to participate. The Trial Outcomes for Massage: Caregiver-Assisted vs. Therapist-Treated (TOMCATT) Study will be a 2-arm, parallel group, randomized clinical trial. Eligible participants will be randomized to one of two study arms: 1) Patients in the therapist-treated arm will receive 3 months of twice weekly massage delivered by certified massage therapists. The second and comparator arm will be a waitlist control. The trial will last 6 months and compare therapist-delivered massage to control on neck pain outcomes. The investigators will compare changes in pain-related disability (primary outcome) between the two groups (Aim 1) and examine secondary outcomes: pain severity, quality of life, depression, anxiety, and stress (Aim 2) as well as exploratory outcomes. To examine the implementation potential of the intervention, including facilitators and barriers, the investigators will conduct post-study, in-depth qualitative interviews of a subsample of study participants (Veteran patients and caregivers) the massage group and the no-longer enrolling CAM group(Aim 3). Lastly, the investigators will assess treatment fidelity and compare the relative intervention costs and budget impact for both interventions. The intervention period will last for 3 months, after which time Veterans will be followed for an additional 3 months.

Innovation: The TOMCATT Study is a novel extension of the investigators' prior work, has strong implementation potential, and innovates by placing caregivers in a treatment delivery role that has the potential to reach a greater number of Veterans with chronic neck pain while also producing substantial cost-savings. Although studies have shown that massage is effective for pain, caregiver-delivered strategies have not been tested or implemented in any systematic way across VA.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain for 6 months or longer
* Neck pain of at least moderate severity (NDI score greater than or equal to 10)

Exclusion Criteria:

* Neck pain secondary to vertebral fracture or metastatic cancer
* Complex neck pain (e.g. cervical radiculopathy or recent whiplash injury)
* Any massage professional massage therapy within the last 6 months
* Active suicidal ideation
* Moderate to severe cognitive impairment
* Pending neck surgery
* Involvement in active pain or massage trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Bair, MD MS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munk N, Daggy JK, Evans E, Kline M, Slaven JE, Laws B, Foote T, Matthias MS, Bair MJ. Therapist-Delivered Versus Care Ally-Assisted Massage for Veterans With Chronic Neck Pain: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 27;11(9):e38950. doi: 10.2196/38950. PMID 36166287
- [Derived] Munk N, Daggy JK, Slaven JE, Foote T, Garner M, Evans E, Laws BV, Matthias MS, Bair MJ. Therapist delivered massage for Veterans with chronic neck pain: a randomized control trial. Pain Med. 2026 Feb 1;27(2):160-169. doi: 10.1093/pm/pnaf118. PMID 40875586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 395 participants were enrolled but 102 randomized to CA-M and not included in the final analysis. Due to high attrition in CA-M (62/98, 63.2%), TOMCATT was modified into a two-arm study (TT-M, WL-C). Three participants were withdrawn post-randomization: one consent revoked and two COVID re-randomizations.
Groups:
- Care Ally Assisted Massage (CA-M): CA-M consisted of in-person training for veteran/care-ally dyads to learn a standardized 30-minue massage routine, instructional DVD, and printed treatment manual. Participants were to complete three care ally-assisted massage sessions weekly for 12-weeks. Outcomes collected at baseline, 1-, 3-, and 6- months included validated measures of neck pain severity and associated disability.
Period: Overall Study
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Started | 145 | 145 | 102
1 Month | 109 | 114 | 43
3 Month | 87 | 109 | 34
6 Month | 77 | 83 | 39
Completed | 77 | 83 | 39
Not Completed | 68 | 62 | 63
Not completed — Lost to Follow-up | 60 | 54 | 17
Not completed — Uncollected | 8 | 8 | 0
Not completed — Ally Health | 0 | 0 | 3
Not completed — Disinterest | 0 | 0 | 22
Not completed — Veteran Health | 0 | 0 | 8
Not completed — Moved | 0 | 0 | 1
Not completed — Scheduling Conflicts | 0 | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Care Ally Assisted Massage: CA-M consisted of in-person training for veteran/care-ally dyads to learn a standardized 30-minue massage routine, instructional DVD, and printed treatment manual. Participants were to complete three care ally-assisted massage sessions weekly for 12-weeks. Outcomes collected at baseline, 1-, 3-, and 6- months included validated measures of neck pain severity and associated disability.
- Total: Total of all reporting groups
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage | Total
Number analyzed (Participants) | 145 | 145 | 102 | 392
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (13.7) | 56.0 (13.7) | 57.2 (14.3) | 55.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 15 | 57
  Male | 125 | 123 | 87 | 335
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 1 | 13
  Not Hispanic or Latino | 137 | 141 | 101 | 379
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 33 | 33 | 19 | 85
  White | 94 | 103 | 77 | 274
  More than one race | 10 | 6 | 3 | 19
  Unknown or Not Reported | 8 | 3 | 3 | 14
Education [Count of Participants; unit: Participants]
  High School Education or Less | 28 | 27 | 22 | 77
  Tech/Business/Associates | 57 | 66 | 45 | 168
  Bachelors or Greater | 49 | 48 | 32 | 129
  Unknown or Not Reported | 11 | 4 | 3 | 18
Marital Status [Count of Participants; unit: Participants]
  Married or Partnered | 84 | 88 | 77 | 249
  Non-Partnered | 51 | 52 | 23 | 126
  Unknown or Not Reported | 10 | 5 | 2 | 17
Employment [Count of Participants; unit: Participants]
  Employed | 69 | 59 | 44 | 172
  Retired | 42 | 50 | 38 | 130
  Unable to Work | 14 | 18 | 8 | 40
  Other | 11 | 13 | 9 | 33
  Unknown or Not Reported | 9 | 5 | 3 | 17
Income [Count of Participants; unit: Participants]
  Comfortable | 77 | 70 | 57 | 204
  Just Enough | 48 | 53 | 34 | 135
  Not Enough | 11 | 14 | 5 | 30
  Don't Know/Refuse to Answer | 1 | 5 | 3 | 9
  Unknown or Not Reported | 8 | 3 | 3 | 14
PTSD Screener [Count of Participants; unit: Participants]
  PTSD Screen Positive | 58 | 54 | 36 | 148
  PTSD Screen Negative | 87 | 91 | 66 | 244
Comorbidity [Median (Full Range); unit: Number of Comorbid Conditions] | 3 [0 to 8] | 3 [0 to 8] | 0 [0 to 0] | 3 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Neck Disability Index
Description: The NDI is the standard instrument for measuring self-rated disability due to neck pain. The NDI was developed as a modification of the well-validated Oswestry Low Back Pain Disability Index. The NDI consists of 10-items that assess pain and functioning. All items are framed as a "problem right now" and are scored on a 6-point numeric rating scores of 0 to 5, with 5 being "worst." The total score ranges from 0 to 50, with higher scores representing greater disability from chronic neck pain. The NDI has strong internal consistency (Cronbach's alpha = 0.80) and construct validity. Scoring of the NDI involves: 1) summing the score for each item (raw score); or 2) raw score can be multiplied by 2 to produce a percentage score. The following scoring intervals aid interpretation: 0 - 4 = no disability; 5 - 14 = mild; 15 - 24 = moderate; 25 - 34 = severe; and > 34 = complete disability. At least a 5-point change is defined as "clinically meaningful."
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 145 | 145 | 102
units on a scale | 20.3 (7.7) | 20.5 (8.5) | 18.3 (7.9)

2. Primary Outcome: Neck Disability Index
Description: as for outcome 1
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 109 | 114 | 43
units on a scale | 18.7 (8.4) | 21.1 (9.2) | 18.1 (8.5)

3. Primary Outcome: Neck Disability Index
Description: as for outcome 1
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 87 | 109 | 34
units on a scale | 17.0 (18.6) | 21.2 (9.0) | 15.1 (8.7)

4. Primary Outcome: Neck Disability Index
Description: as for outcome 1
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 77 | 83 | 39
units on a scale | 18.5 (8.3) | 21.6 (9.8) | 14.9 (8.3)

5. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory is an 11-item, multidimensional pain measurement tool with reliability in patients with arthritis as well as other pain conditions. The BPI rates the intensity of pain as well as the interference of pain with mood, physical activity, work, social activity, relations, sleep, and enjoyment of life. The BPI has a score range from 0-10 with higher scores representing more severe pain and more pain interference.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 145 | 145 | 102
units on a scale | 6.1 (1.7) | 6.2 (1.8) | 6.0 (1.9)

6. Secondary Outcome: Medical Outcomes Study Veterans RAND 36 Item Health Survey (VR-36) (Modified From Medical Outcomes Study SF-36)
Description: Health-related quality of life will be measured with the VR-36, a modified version of the Medical Outcomes Study SF-36 widely used in VA research and available in the public domain. Internal consistency is high. The VR-36 is scored 0-100 with higher scores representing improved health related quality of life.
Time Frame: Baseline
Population: Participants refused to answer items from this instrument.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage
Number analyzed (Participants) | 144 | 142 | 95
units on a scale | 45.7 (13.3) | 46.2 (14.2) | 47.0 (12.3)

7. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 5
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 109 | 114 | 42
units on a scale | 5.1 (1.9) | 6.0 (2.0) | 5.5 (1.7)

8. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 5
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 87 | 109 | 34
units on a scale | 4.5 (2.0) | 6.0 (1.9) | 4.6 (2.1)

9. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 5
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage (CA-M)
Number analyzed (Participants) | 77 | 83 | 37
units on a scale | 4.7 (2.2) | 5.7 (1.9) | 4.5 (2.4)

10. Secondary Outcome: Medical Outcomes Study Veterans RAND 36 Item Health Survey (VR-36) (Modified From Medical Outcomes Study SF-36)
Description: as for outcome 6
Time Frame: 1 Month
Population: Participants refused to answer items from this instrument.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage
Number analyzed (Participants) | 107 | 108 | 42
units on a scale | 47.4 (13.4) | 46.7 (14.2) | 47.7 (13.2)

11. Secondary Outcome: Medical Outcomes Study Veterans RAND 36 Item Health Survey (VR-36) (Modified From Medical Outcomes Study SF-36)
Description: as for outcome 6
Time Frame: 3 Month
Population: Participants refused to answer items from this instrument.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage
Number analyzed (Participants) | 87 | 105 | 34
units on a scale | 47.9 (12.0) | 45.7 (14.4) | 51.3 (15.0)

12. Secondary Outcome: Medical Outcomes Study Veterans RAND 36 Item Health Survey (VR-36) (Modified From Medical Outcomes Study SF-36)
Description: as for outcome 6
Time Frame: 6 Month
Population: Participants refused to answer items from this instrument.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage
Number analyzed (Participants) | 77 | 83 | 38
units on a scale | 45.8 (12.8) | 43.4 (15.8) | 49.7 (11.8)

ADVERSE EVENTS:
Time Frame: SAEs, AEs, and UAPs were collected from the time of study entry until the end of study participation, an average of 6 months.
Arm/Group | Therapist Treated Massage (TT-M) | Wait List Control (WL-C) | Care Ally Assisted Massage
All-Cause Mortality (participants affected / at risk) | 1/145 | 0/145 | 1/102
Serious Adverse Events (participants affected / at risk) | 10/145 | 3/145 | 6/102
Other Adverse Events (participants affected / at risk) | 106/145 | 13/145 | 14/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapist Treated Massage (TT-M) (N=145) | Wait List Control (WL-C) (N=145) | Care Ally Assisted Massage (N=102)
DEATH (Nervous system disorders) | 1 | 0 | 1
PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
INPATIENT ADMISSION (Nervous system disorders) | 1 | 1 | 0
SURGERY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
PAIN (Nervous system disorders) | 1 | 0 | 0
SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SURGERY (Surgical and medical procedures) | 2 | 0 | 0
INPATIENT ADMISSION (Infections and infestations) | 0 | 1 | 0
INPATIENT ADMISSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PAIN (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapist Treated Massage (TT-M) (N=145) | Wait List Control (WL-C) (N=145) | Care Ally Assisted Massage (N=102)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1
HEADACHE (Nervous system disorders) | 3 | 1 | 0
INFECTION (Infections and infestations) | 4 | 2 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 5 | 0
SORENESS (Musculoskeletal and connective tissue disorders) | 31 | 1 | 1
STIFFNESS (Musculoskeletal and connective tissue disorders) | 18 | 2 | 0
SURGERY (Surgical and medical procedures) | 3 | 1 | 2
DISCOMFORT (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
SHOULDER DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
DIZZINESS (General disorders) | 3 | 0 | 1
HEART PAIN (Cardiac disorders) | 1 | 0 | 0
LEG PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
NUMBNESS (Nervous system disorders) | 1 | 0 | 0
PAIN (Musculoskeletal and connective tissue disorders) | 12 | 0 | 2
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
STOMACH ISSUES (Gastrointestinal disorders) | 1 | 0 | 0
TENDERNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SHOULDER PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
HYPERVENTILATING (Psychiatric disorders) | 0 | 0 | 1
KIDNEY LUMPS (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT03100539/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT03100539/ICF_001.pdf